CLINICAL TRIAL: NCT06827925
Title: Exploring the Effectiveness of Flipped Education in Distance Digital Learning for Long-term Care Nurses on Pressure Injury Staging Interpretation
Brief Title: Telemedicine Wounds
Acronym: Staging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Collaborators: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WYMeiYu2025
Record Dates: First submitted 2025-01-13; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Pressure Injury
Keywords: Long-term care; nurse; Telemedicine; pressure injury; staging Interpretation
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- routine (No Intervention): Not receiving Distance Digital Learning of Flipped Education
- Distance Digital Learning (Active Comparator): Distance Digital Learning
  Interventions: Other: Distance Digital Learning

INTERVENTIONS:
Other: Distance Digital Learning — receiving Distance Digital Learning of Flipped Education
  Arms: Distance Digital Learning

SUMMARY:
This study aims to explore the effectiveness of the flipped education model applied to distance digital learning in enhancing the pressure injury staging interpretation skills of long-term care nursing staff. A quasi-experimental design was employed, dividing participants into a flipped education group and a conventional digital learning group. Pre- and post-intervention assessments were conducted to evaluate knowledge and skills, and differences in satisfaction and cognitive load were compared.

ELIGIBILITY:
Inclusion Criteria:

* Home care worker
* Those who have access to a smartphone and the Internet
* After the purpose of the study was explained, they agreed to participate in the study and signed the consent form.

Exclusion Criteria:

* Business managers or administrative managers who do not actually provide frontline care at the patient's home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure injury staging interpretation test | One month before intervention， and one month after intervention
  The scale consists of 21 questions and the assessment takes approximately 10 to 12 minutes. A correct answer will earn 1 point, and an incorrect answer will earn 0 points. The total score ranges from 0 to 21, and the calculation method is {(number of correct answers/21 questions)*100%} as the test score, rounded to the first decimal place. Higher scores represent better knowledge of the degree of crush injury interpretation.

SECONDARY OUTCOMES:
Satisfaction with teaching mode | One month before intervention， and one month after intervention
  It is a structured questionnaire with 10 questions in total, focusing on teaching objectives, teaching content design, multimedia design, and self-conscious learning outcomes. The ratings were given on a five-point Likert scale, ranging from 5 (very satisfied), 3 (no opinion), to 1 (very dissatisfied). The total score ranges from 10 to 50, with higher scores indicating greater satisfaction with the educational strategy for pressure injury care and management.
Cognitive load of learning | One month before intervention， and one month after intervention
  The cognitive load scale assesses the subjective feelings of the subjects during the learning process and can be divided into two subscales: external cognitive load and augmentative cognitive load. The questionnaire consists of 5 questions, using a five-point Likert scale ranging from "strongly agree" (1 point) to "strongly disagree" (5 points). Total scores range from 5 to 25, with higher extrinsic cognitive load scores indicating lower cognitive load and lower accretive cognitive load scores indicating higher accretive cognitive load.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University, Taichung, Taiwan, Taiwan